CLINICAL TRIAL: NCT02521571
Title: The Resilience Alliance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 12-00568
Record Dates: First submitted 2015-08-07; First posted 2015-08-13 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Secondary Traumatic Stress
MeSH Terms: conditions — Compassion Fatigue

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Behavioral: Resiliance Alliance
- Control Group (Placebo Comparator)
  Interventions: Behavioral: Secondary traumatic stress training

INTERVENTIONS:
Behavioral: Resiliance Alliance — The intervention is 6 months long & is delivered through weekly sessions held in the participating child protective offices. The sessions follow a 4-week cycle with the participants changing each week of the cycle: (1) CPS alone, by units; (2) CPS/Supervisor units; (3) Child Protective Manager and CPS/Supervisor units; and (4) CPSs & Supervisors/Managers separately.
  Participating staff are introduced to a resilience-related topic or skill, and receive a brief didactic training on that topic. Staff then engage in a group activity, which is designed to help them apply the new topic or skill to the workplace. Each module wraps up with a relaxation or exercise to help staff transition back into their work responsibilities; the facilitator can pick among the selection provided based on their sense of what would be helpful for the group. Staff are also given handouts and activities to do during the week.
  Arms: Intervention Group
Behavioral: Secondary traumatic stress training — These trainings will take place in two parts (for a total of 3 hours) and include an overview of secondary traumatic stress and its impact on child welfare staff, and some strategies staff can use to protect themselves from STS - essentially a "summary" version of what the intervention group will receive over the 24 weeks of the intervention. The investigators consider this training to represent "treatment as usual," as from our experience it is often how child welfare agencies address the issue of secondary traumatic stress among their staff.
  Arms: Control Group

SUMMARY:
The Resilience Alliance is a skill-based staff development intervention for child protective staff that focuses on improving job satisfaction, resilience, optimism and social support, while decreasing attrition, stress reactivity and burnout. The investigators believe that the intervention will enhance the capacity of child welfare workers to care for themselves, which will result in them providing better care for the children and families involved with the child welfare system.

The Resiliance Alliance will be implemented in two child protective offices, Manhattan Zone C and Brooklyn Zone B. Staff from two additional offices (Staten Island Zone A and Brooklyn Zone C) will serve as a control group. A web-based survey will be administered in the group receiving the Resiliance Alliance intervention prior to intervention, at completion of the intervention, and 3 months post completion. The control group will be given a two-part training (3 hours in total) on secondary traumatic stress. The control group will then be asked to complete the same survey as the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Administration for Children's Services (ACS) employees working at one of four offices: Manhattan Zone C, Brooklyn Zone B, Staten Island Zone A and Brooklyn Zone C
* Adults aged 18 years or older
* English-speaking

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2011-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change in Survey Over Time | At baseline, upon conclusion of the intervention (6 months), and 3 months post-intervention
  The survey results will be compared between the two groups at three different timepoints as listed above

CONTACTS AND LOCATIONS:
Overall Officials: Claude Chemtob, Principal Investigator — NYU MEDICAL CENTER
Locations (4):
- United States (4):
  - Brooklyn ACS Borough Office, Brooklyn, New York
  - Manhattan ACS Borough Office, New York, New York
  - Staten Island ACS Borough Office, Staten Island, New York
  - Bronx ACS Borough Office, The Bronx, New York